CLINICAL TRIAL: NCT03971201
Title: A Randomized Phase II Trial of Surgery Plus Sorafenib vs. Sorafenib Alone for Hepatocellular Cancer (HCC) With Portal Vein Invasion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: White Plains Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); Sun Yat-sen University (Other); West China Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Anhui Provincial Hospital (Other Government); Fujian Cancer Hospital (Other Government); Wenzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190507
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Cancer
Keywords: portal vein invasion
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Surgery plus sorafenib (Experimental): surgical resection followed by adjuvant sorafenib
  Interventions: Procedure: hepatic resection; Drug: Sorafenib
- sorafenib only (Active Comparator): sorafenib only
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Procedure: hepatic resection — removal of portion of liver containing cancer
  Arms: Surgery plus sorafenib
Drug: Sorafenib — sorafenib either as adjuvant therapy after resection or as only treatment

SUMMARY:
Patients with HCC with portal vein involvement not involving the bifurcation (vP1-vP3) and no evidence of extra-hepatic spread will be enrolled. Patients will be required to have Child's A liver function and no significant portal hypertension. Patients will be randomly assigned with a 1:1 ratio to either surgery followed by adjuvant sorafenib or sorafenib alone. Patients will be followed by serial imaging. The primary end-point is overall survival.

DETAILED DESCRIPTION:
Trial design

Surgery + sorafenib vs. sorafenib 100 patients per arm Centralized randomization by CRO Need to call CRO for treatment allocation Primary end-point - OS Secondary end-point Progression free survival (PFS) Randomized 1:1 Stratification Vp1-2 vs. Vp3 AFP ≤400 vs AFP >400 Intention to treat Surgery aborted or R1-2 resection will remain in surgical arm No cross over CT scan chest/abdomen 4 weeks after surgery as post-operative baseline Will not alter treatment allocation Will allow for PFS measurement in surgical arm CT scan chest/abdomen pelvis Q 12 weeks after initiation sorafenib Patients progressing on sorafenib allowed 2nd line treatment Regorafenib or lenvatinib - if approved in China Dose reduction sorafenib as per protocol

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of HCC A) 1st diagnosis of HCC - no prior treatments of HCC B) Diagnosis made by contrast enhanced CT or MRI with arterial and portal phases

1. Arterial enhancement
2. Venous washout
3. Expanding/enhancing tumor thrombus seen in portal vein Extent of HCC spread A) Vp1-3 (Japanese system) - VP1-2 (Cheng criteria - Shanghai) B) No involvement of main portal vein Vp4 (Japanese system) - Vp3 Shanghai C) No evidence of extra-hepatic spread in abdomen D) No evidence of hepatic vein or vena cava invasion Need for Biopsy A) Patients not meeting above criteria B) Absence of underlying liver disease Demographics A) Age ≥ 18 Women of reproductive age A) Negative pregnancy test B) Must be on birth control for duration of study Able to provide informed consent No prior malignancy A) Excluding basal/squamous cell skin cancers B) Excluding superficial bladder cancer C) Excluding cervical cancer Underlying liver disease A) HBV, HCV, alcohol, or none B) All HBV patients must be placed on anti-viral therapy prior to any treatment and continue through entire study C) Co-infection HBV with HCV excluded D) HIV infection excluded Liver function/Performance status A) Child's A or B7 liver function B) Absence of clinical portal hypertension

a. Platelet count ≥ 100,000 b. No evidence of varices or splenomegaly on imaging c. No ascites ECOG performance status 0-1 Tumor characteristics A) Size of largest tumor ≤ 10cm B) <50% of liver volume involved by tumor C) Multiple tumors allowed D) All tumors all confined to same lobe as PV involvement E) Hepatic Vein or Inferior Vena Cava involvement excluded Non-contrast CT of chest A) No lung metastases B) Involvement of gallbladder and diaphragm allowed C) Involvement of omentum allowed D) Involvement of abdominal wall allowed E) Involvement of colon, stomach, duodenum excluded

Exclusion Criteria:

Unable to provide informed consent Age <18 years Unable to take anti-viral medication for hepatitis B Unable to take sorafenib Medically unfit for surgery Prior malignancy other than those specifically allowed by study Prior treatment of HCC Tumor characteristics A) HCC >10cm B) Bilobar tumor C) Mixed cholangiocarcinoma HCC D) Extra-hepatic tumor E) Tumor involving stomach, duodenum or colon F) Tumor involving hepatic veins or vena cava G) Tumor involving portal vein bifurcation

Liver disease A) Liver function decompensated beyond Child's B7 B) Significant portal hypertension - splenomegaly, varices, ascites or platelet count <100,000 C) Co-infection with HBV and HCV D) Co-infection with HIV ECOG performance status >1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2-3 year
  time from randomization to death

SECONDARY OUTCOMES:
progression free survival | 3-12 months
  time from initiation of intervention until progression as defined by RESIST

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Data will not be shared